CLINICAL TRIAL: NCT01626703
Title: Effect of Depressin Screening and Care Program at Community Health Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Clinical Research Coordination Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Hyeon Woo Yim, professor, National Clinical Research Coordination Center, Seoul, Korea
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: A102065_2012_2
Record Dates: First submitted 2012-06-20; First posted 2012-06-25 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Depression; Screening; Elderly
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- intervention (Experimental): remiding call
  Interventions: Other: Reminding call
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Reminding call
  Arms: intervention

SUMMARY:
Depression affect between 5% and 10% of older adults seen in the primary care setting.Late-life depression is often chronic or recurrent and is associated with substantial suffering, functional impairment, and diminished health-related quality of life.Depressed, older primary care patients are frequent users of general medical services and may have poor adherence to medical treatments.They are also at increased risk of death from suicide and medical illnesses. The aim of this study is to examine whether depression screening and health care practitioner feedback are increased depression treatment rate.

Depression screening is provided 60 or more who visited community health care center with a 15-item Geriatric Depression Scale.GDS scores of 10 or more were classified depression positive. Intervention group participants received twice remind calls from primary care nurse.

ELIGIBILITY:
Inclusion Criteria:

* 60 or more
* 10 or more in GDS scor

Exclusion Criteria:

* severe cognitive problem

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Reuptake rate | 12 weeks

SECONDARY OUTCOMES:
reduced depressive symptoms | 12 weeks
  Geriatric Depression Scale Short Form (SGDS)
changed perceived heath status | 12 weeks
  Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Chungju community health care center, Chungju, Choongbuk, South Korea